CLINICAL TRIAL: NCT02638480
Title: A Prospective Randomized Trial to Examine the Effectiveness of KneeMD on Flexion Contracture in Total Knee Arthroplasty Patients
Brief Title: Effectiveness of KneeMD on Flexion Contracture in Total Knee Arthroplasty Patients
Acronym: KneeMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anne Arundel Health System Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 811229
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Flexion Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control subjects will be treated with only the current SOC including NSAIDs and physical therapy.
- Experimental (Experimental): The experimental subjects will be treated with current SOC and will also use a kneeMD splint 3 times a day for 20 minutes per session
  Interventions: Device: KneeMD

INTERVENTIONS:
Device: KneeMD — KneeMD is a subject-controlled knee rehabilita¬tion device that helps subjects who have undergone total knee replacements or other major knee surger¬ies improve range of motion and stretch in extension.
  Arms: Experimental

SUMMARY:
The purpose of this study is to evaluate the effect of the KneeMD subject-controlled knee rehabilitation device on the incidence of postoperative flexion contracture.

DETAILED DESCRIPTION:
Postoperative flexion contracture (FC), defined as >10°, is the most common disabling early complication of primary total knee replacement (TKR) surgery, affecting up to 6% of all subjects. A knee flexion of 65° is required to walk, 70° is needed to lift an object from the floor, 85° to climb stairs, 95° for optimal sitting and standing, and 105° to tie shoelaces. With growing subject and physician expectations for function and range of motion (ROM) after surgery, FC complications have become an early measure of success in TKR surgery.

The purpose of this study is to evaluate the effect of the KneeMD subject-controlled knee rehabilitation device on the incidence of postoperative FC. The primary endpoints are the preoperative change in active range of motion (AROM) and the incidence of postoperative FC at 2 weeks. Secondary endpoints include the change in AROM in subjects with postoperative FC.

ELIGIBILITY:
Inclusion Criteria:

1. Measurable Knee Flexion Contracture, with deficit limiting Active Range of Motion (AROM) and Passive Range of Motion (PROM) by at least - 10°
2. 18 years of age and older
3. Able to understand informed consent and willingness to conform to trial responsibilities

Exclusion Criteria:

1. Previous surgical treatment of knee, including tibial osteotomy
2. Botulinum Toxin Treatment within the last four months
3. Mechanical joint impingement
4. Neuromuscular pathologies such as epilepsy
5. Treatment with quinolone, antibiotic medication
6. Pregnant or nursing
7. Fractures
8. Osteomyelitis or any orthopedic infection
9. Extensor mechanism dysfunction
10. Knee joint neuropathy
11. Previous Stroke or Brain Injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
AROM | 4 weeks after randomization
  Change in maximal active range of motion in

SECONDARY OUTCOMES:
AROM | 2 weeks postoperatively
  Active Range of motion in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Arundel Medical Center, Annapolis, Maryland, United States

REFERENCES:
- [Background] Gonzalez Della Valle A, Leali A, Haas S. Etiology and surgical interventions for stiff total knee replacements. HSS J. 2007 Sep;3(2):182-9. doi: 10.1007/s11420-007-9053-4. PMID 18751792
- [Background] Pariente GM, Lombardi AV Jr, Berend KR, Mallory TH, Adams JB. Manipulation with prolonged epidural analgesia for treatment of TKA complicated by arthrofibrosis. Surg Technol Int. 2006;15:221-4. PMID 17029180
- [Background] Yercan HS, Sugun TS, Bussiere C, Ait Si Selmi T, Davies A, Neyret P. Stiffness after total knee arthroplasty: prevalence, management and outcomes. Knee. 2006 Mar;13(2):111-7. doi: 10.1016/j.knee.2005.10.001. Epub 2006 Feb 20. PMID 16490357
- [Background] Laubenthal KN, Smidt GL, Kettelkamp DB. A quantitative analysis of knee motion during activities of daily living. Phys Ther. 1972 Jan;52(1):34-43. doi: 10.1093/ptj/52.1.34. No abstract available. PMID 5061683
- [Background] Schurman DJ, Parker JN, Ornstein D. Total condylar knee replacement. A study of factors influencing range of motion as late as two years after arthroplasty. J Bone Joint Surg Am. 1985 Sep;67(7):1006-14. PMID 4030819
- [Background] Mitsuyasu H, Matsuda S, Miura H, Okazaki K, Fukagawa S, Iwamoto Y. Flexion contracture persists if the contracture is more than 15 degrees at 3 months after total knee arthroplasty. J Arthroplasty. 2011 Jun;26(4):639-43. doi: 10.1016/j.arth.2010.04.023. Epub 2010 Jun 11. PMID 20541887
- [Background] Ritter MA, Lutgring JD, Davis KE, Berend ME, Pierson JL, Meneghini RM. The role of flexion contracture on outcomes in primary total knee arthroplasty. J Arthroplasty. 2007 Dec;22(8):1092-6. doi: 10.1016/j.arth.2006.11.009. PMID 18078875
- [Background] Goudie ST, Deakin AH, Ahmad A, Maheshwari R, Picard F. Flexion contracture following primary total knee arthroplasty: risk factors and outcomes. Orthopedics. 2011 Dec 6;34(12):e855-9. doi: 10.3928/01477447-20111021-18. PMID 22146201
- [Background] Aderinto J, Brenkel IJ, Chan P. Natural history of fixed flexion deformity following total knee replacement: a prospective five-year study. J Bone Joint Surg Br. 2005 Jul;87(7):934-6. doi: 10.1302/0301-620X.87B7.15586. PMID 15972905
- [Background] Lam LO, Swift S, Shakespeare D. Fixed flexion deformity and flexion after knee arthroplasty. What happens in the first 12 months after surgery and can a poor outcome be predicted? Knee. 2003 Jun;10(2):181-5. doi: 10.1016/s0968-0160(02)00102-3. PMID 12788004
- [Background] Koh IJ, Chang CB, Kang YG, Seong SC, Kim TK. Incidence, predictors, and effects of residual flexion contracture on clinical outcomes of total knee arthroplasty. J Arthroplasty. 2013 Apr;28(4):585-90. doi: 10.1016/j.arth.2012.07.014. Epub 2012 Nov 8. PMID 23142447